CLINICAL TRIAL: NCT04837248
Title: Design and Evaluation of the Effects of a Physical Therapy Program With Digital Support in Patients With Breast Cancer Surgery. A Clinical Trial.
Brief Title: Design and Evaluation of the Effects of a Physical Therapy Program With Digital Support in Patients With Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacion para la Investigacion Biomedica del Hospital Universitario Ramon y Cajal (Other)
Responsible Party: Principal Investigator, Ana Belén Romojaro Rodríguez, Physiotherapist, Fundacion para la Investigacion Biomedica del Hospital Universitario Ramon y Cajal
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PI-2021-3
Record Dates: First submitted 2021-04-06; First posted 2021-04-08 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Breast Cancer
Keywords: Exercise; Muscle Weakness; Lymphedema; Fatigue; Depression
MeSH Terms: conditions — Breast Neoplasms; Motor Activity; Muscle Weakness; Lymphedema; Fatigue; Depression

STUDY DESIGN:
Intervention Model Description: Group 1. Conventional treatment. Patients will be treated by means of a physiotherapy programme without digital support. They will be given a written document with exercises and recommendations on the first day.
  Group 2. Experimental treatment. Patients will be treated with a digitally supported physiotherapy programme.
Who Masked: Outcomes Assessor
Masking Description: The assessor will assess patients at baseline, 6 weeks, 12 weeks, and 6 months and will not know which arm of the study each patient belongs to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1. Conventional treatment (Active Comparator): Patients will be treated with a physiotherapy programme without digital support.
  Interventions: Other: Active Comparator: Group 1. Conventional treatment
- Group 2. Experimental treatment. (Experimental): Patients will be treated using a digitally supported physiotherapy programme.
  Interventions: Other: Experimental: Group 2. Experimental treatment.

INTERVENTIONS:
Other: Active Comparator: Group 1. Conventional treatment — Patients will be treated using a physiotherapy programme without digital support. A written document with exercises and recommendations will be given to them on the first day. This booklet will detail the exercises they can do depending on their surgery and the weeks elapsed, as well as the recommendations adapted according to the needs identified in the motivational interview (MI). This is the treatment that is currently being applied in the hospital.
  The patient will carry out the treatment at home and will come back after 20 sessions for the corresponding assessment.
  Arms: Group 1. Conventional treatment
Other: Experimental: Group 2. Experimental treatment. — A digitally supported physiotherapy programme including:
  * Group session: expectations, interests, experiences with regard to their health problem and the consequences on their life, joint exercise and discussion with subsequent debate will be held.
  * Exercise session: each week, patients will find different exercise videos on the platform according to the phase of recovery in which each one of them is, having been previously evaluated in the group session.
  * Relaxation session: this will be carried out by means of audio that will be posted on the platform and that the patient will be able to perform simultaneously.
  * Empowerment session: audio sessions that will deal with those needs that frequently arise after breast surgery in their daily lives, focusing on limiting beliefs (e.g. fear of moving), positive thoughts and information extracted from the motivational interview that should be developed.
  Arms: Group 2. Experimental treatment.

SUMMARY:
Breast cancer surgery usually results in reduced range of motion of the shoulder joint, weakness of the musculature and altered scapular kinematics during movement. These factors limit activities of daily living, so rehabilitation exercises help to restore function after shoulder surgery.

Women with breast cancer often have a life conditioned by the sequelae or morbidity secondary to the treatment of the disease and, despite the high cure rate, many patients are unable to regain their initial quality of life. Cancer therapies can leave physical, psychological and psychosocial sequelae, which may manifest themselves or persist even years after the end of treatment.

For all these reasons, patients who have undergone cancer treatment need physical rehabilitation as well as psychological and social care to support them in their new stage of life, and to optimise the rehabilitation programme, it is necessary to identify each patient's individual needs,

The digital support proposed in this study enables the development of a physiotherapy programme for patients with breast cancer in a situation of health crisis, which includes providing assistance, information, accompaniment, help and treatment to these patients in a comprehensive way, based on the biopsychosocial model.

DETAILED DESCRIPTION:
DESIGN: Single-centre, assessor-blinded, parallel-group, randomised controlled clinical trial.

METHODS: The study will be carried out at the Ramon y Cajal hospital with 92 patients diagnosed and operated on for breast cancer.

Patients who come to the consultation of the rehabilitation doctors will be assessed, considering the inclusion and exclusion criteria. Those who may be candidates will be informed about the study and referred to the physiotherapy department where the treatment orders for these patients will be received and an appointment will be made. This is the start of the recruitment phase.

Those who meet the criteria and agree to participate in the study will be assigned an identification code and will be randomised into the two groups, the intervention group and the conventional treatment group.

Patients who do not meet the inclusion criteria or refuse to participate in the study will receive conventional treatment.

A 6-month pilot study will be conducted to better define patient identification, inclusion criteria, recruitment and adjustment of the intervention if required.

Once the pilot study is completed, the intervention clinical trial will begin. A first analysis of all variables will be performed after the intervention phase of the trial, 6 weeks after inclusion in the study.

An interim analysis will also be performed at 3 months in which the same variables as at 6 weeks will be assessed. This will be the main analysis of the study.

The final analysis will be carried out 6 months after inclusion in the study, and this will conclude the follow-up phase.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of stage I, II or III of Breast cancer treated by surgery.
* Medical authorisation for participation.
* Internet access.
* Basic computer skills.
* Signed informed consent.
* No bilateral mastectomy.
* No metastases.
* Post-intervention period of 10 days to 3 months.
* Age 18-85 years.
* No previous shoulder pathologies.
* No pathology that prevents exercise.
* Understanding of the Spanish language.

Exclusion Criteria:

* Breast cancer treated without surgery.
* Patient in severe psychiatric treatment who may present difficulties for participation in the study.
* Stage IV cancer.
* Any other clinical condition or previous therapy that contraindicates one or more of the techniques included in the programme, as the intervention may not be safe for the patient and therefore the person would not be eligible to participate in the study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2021-08-02 (Actual); Primary Completion 2024-10-28 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Disabilities of the Arm, Shoulder and Hand Score (DASH) | 12 weeks
  Global assessment of the functionality of the upper limb,
Disabilities of the Arm, Shoulder and Hand Score (DASH) | 3 months
  Global assessment of the functionality of the upper limb,

SECONDARY OUTCOMES:
European organization for research and treatment of cancer quality life questionnaire core 30. (QLQ-C30-B23) | 12 weeks
  Questionnaire to assess quality of life in cancer patients. Module B23, which is specific to breast cancer, will be used.
Range Of Motion (ROM) | 12 weeks
  Goniometry of joint range
Tampa Scale for Kinesiophobia (TSK-11SV) | 12 weeks
  The TSK is an 11-item self-report measure related to fear of movement and re-injury from movement.
Brief Pain Inventory (BPI) | 12 weeks
  The BPI is a multidimensional pain assessment tool that provides information on pain intensity and its interference with patients' daily activities. It also assesses the description, the location of pain and the level of relief provided by the treatment.
Hospital Anxiety and Depression Scale (HADS) | 12 weeks
  Questionnaire to measure levels of anxiety and depression in these people.

CONTACTS AND LOCATIONS:
Locations (1):
- Fundacion Hospital Ramón y Cajal, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pellini F, Granuzzo E, Urbani S, Mirandola S, Caldana M, Lombardi D, Fiorio E, Mandara M, Pollini GP. Male Breast Cancer: Surgical and Genetic Features and a Multidisciplinary Management Strategy. Breast Care (Basel). 2020 Feb;15(1):14-20. doi: 10.1159/000501711. Epub 2019 Sep 13. PMID 32231493
- [Background] Hidding JT, Beurskens CH, van der Wees PJ, van Laarhoven HW, Nijhuis-van der Sanden MW. Treatment related impairments in arm and shoulder in patients with breast cancer: a systematic review. PLoS One. 2014 May 9;9(5):e96748. doi: 10.1371/journal.pone.0096748. eCollection 2014. PMID 24816774
- [Background] van Egmond MA, van der Schaaf M, Vredeveld T, Vollenbroek-Hutten MMR, van Berge Henegouwen MI, Klinkenbijl JHG, Engelbert RHH. Effectiveness of physiotherapy with telerehabilitation in surgical patients: a systematic review and meta-analysis. Physiotherapy. 2018 Sep;104(3):277-298. doi: 10.1016/j.physio.2018.04.004. Epub 2018 Jun 19. PMID 30030037